CLINICAL TRIAL: NCT01867788
Title: Ancillary Longitudinal CSF Collection Study in the Harvard Biomarker Study - HBS2
Acronym: HBS2
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH); Harvard Medical School (HMS and HSDM) (Other)
Responsible Party: Principal Investigator, Clemens Scherzer, MD, Associate Professor of Neurology, Brigham and Women's Hospital
Other Study IDs: NS082157; U01NS082157 (NIH)
Record Dates: First submitted 2013-05-30; First posted 2013-06-04 (Estimated); Last update posted 2016-01-12 (Estimated); Status verified 2016-01

CONDITIONS: Parkinson's Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 36 Months
Biospecimen Retention: Samples With DNA — Whole blood, plasma, CSF, RNA, DNA
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Parkinson's disease subjects
- Healthy Control subjects

SUMMARY:
The Harvard Biomarker Study is a Harvard-wide, longitudinal case-control study designed for discovering, replicating, and developing biomarkers for Parkinson's disease and Alzheimer's disease. High-quality biosamples and high-resolution clinical phenotypes are tracked at three visits over a two-year period for more than 2,000 individuals with early-stage PD, MCI/AD, and controls without neurologic disease.

The present "Ancillary Longitudinal CSF Collection Study (short HBS2)" is an ancillary study to the parent Harvard Biomarker Study. HBS2 is funded by the NINDS. In HBS2, 75 participants are more intensely studied and followed over a three-year time period. Clinical data and blood biospecimens are collected every six months and four annual CSF collections are performed. Biospecimens and clinical data are deposited into the NINDS PD Biomarkers Program (PDBP) Repository and the Data Management Resource (DMR) and are accessible through the PDBP DMR website.

ELIGIBILITY:
Inclusion Criteria for Cases with PD:

* Age ≥ 21
* UK Parkinson's Disease Society Brain Bank criteria or movement disorder specialist diagnosis of PD
* Hoehn & Yahr stage ≤ 3.0
* Mini Mental State Exam score >21 OR authorized legal guardian available to sign consent
* Able to provide informed consent

Inclusion Criteria for Controls:

* Age ≥ 21
* Absence of any neurological disease
* No family history of a first-degree relative with PD
* Mini Mental State Exam score >21 OR authorized legal guardian available to sign consent
* Able to provide informed consent

Exclusion Criteria for Cases and Controls:

* Acquired or inherited bleeding disorders
* Hematologic malignancies
* Hematocrit < 30
* Active ulcer or active colitis
* Known pregnancy
* Clinical contraindications to lumbar puncture (including: known mass lesion of the CNS or evidence for raised intracranial pressure on fundoscopic exam; abnormal coagulation tests; platelet count < 50,000; subject on warfarin (coumadin), heparin, dabigatran, rivaroxiban or apixaban; subject on both aspirin and clopidogrel (Plavix); infection near the LP site or spinal deformity; known allergy to lidocaine)

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Two tertiary care centers.
Sampling Method: Non-Probability Sample
Enrollment: 76 (Actual)
Dates: Start 2012-09; Primary Completion 2017-09 (Estimated); Study Completion 2017-09 (Estimated)

PRIMARY OUTCOMES:
Mean difference in the relative abundance of prioritized transcripts measured in CSF in the PD group compared to the healthy control group. | Enrollment visit

CONTACTS AND LOCATIONS:
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States